CLINICAL TRIAL: NCT02987751
Title: A Prospective, Multicentric, Randomized, Open-Label Comparison of a Long-Acting Basal Insulin Analog Glargine Plus Glulisine With Premixed Insulin in Adult Patients With Type 2 Diabetes Mellitus
Brief Title: A Study on Comparison of Glargine Plus Glulisine With Premixed Insulin in Type 2 Diabetes Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDRFARH007
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Insulin Glargine; insulin glulisine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glargine + Glulisine (Experimental): Insulin Glargine + Glulisine (12U/day + 4U/day) at pre-breakfast/dinner for 24 weeks
  Interventions: Drug: Glargine + Glulisine
- Premixed Analogue Insulin (70/30) (Active Comparator): Premixed analogue Insulin (70/30) 16U/day at pre-breakfast/dinner for 24 weeks
  Interventions: Drug: Premixed analogue insulin (70/30)

INTERVENTIONS:
Drug: Glargine + Glulisine — Glargine should be taken 30 minutes before breakfast/dinner, the dose is adjusted as per fasting blood glucose during each visit and Glulisine should be taken 20 minutes before breakfast/dinner, the dose is adjusted as per postprandial blood glucose during each visit
  Other Names: Lantus + Apidra
  Arms: Glargine + Glulisine
Drug: Premixed analogue insulin (70/30) — Premixed analogue insulin should be taken 30 minutes before breakfast/dinner, the dose is adjusted as per fasting blood glucose during each visit.
  Other Names: Novomix
  Arms: Premixed Analogue Insulin (70/30)

SUMMARY:
This study is a multicentre, randomized, open label on comparison of a Long-Acting Basal Insulin Analog Glargine plus Glulisine with Premixed Insulin in Adult Patients with Type 2 Diabetes Mellitus in 200 patients that will be conducted in seven centers in Tamil Nadu. The primary outcome measures will be to compare the change in HbA1c from baseline to week 24 between Glargine OD + Glulisine in comparison with Premixed insulin initiation in insulin naïve patients with T2DM. The secondary outcomes is to compare the following in the two arms between baseline and 24 weeks Fasting plasma glucose, Postprandial glucose, 7-point self-monitored blood glucose (SMBG) profiles, Percentage of participants with HbA1c < 7%, Insulin dose, Overall adverse events, Symptomatic Hypoglycemia, Severe hypoglycemic, Weight, BMI and Blood pressure.

DETAILED DESCRIPTION:
The subjects will be invited to the study centre from the local population who are willing to participate in the trial. Each subject will be informed both orally and in writing about the study prior to inclusion in the study and only the subjects who give written informed consent will be included. The selection of the subjects is based on the inclusion and exclusion criteria defined in the protocol. The selected subjects will be given a screening number and subjected to screening procedure to find out eligible candidates for enrollment. The screening procedure includes obtaining subject's anthropometric data, baseline symptomatology, medical history, vital signs, physical examination, laboratory investigations like blood glucose (fasting & 2hr after meal), HbA1c, Urea, Creatinine, Liver function test, Lipid profile, Urine albumin/creatinine ratio, urine pregnancy (if applicable) and ECG.

This will be followed by 2 weeks run in period for eligible patients to ensure patients are on stable dose of oral therapy and Metformin not < 1500 mg/day. Sulfonylurea will be stopped.

All the eligible patients as per the inclusion criteria (HbA1c ≥7.5% to ≤ 10.5%, fasting blood glucose ≥ 150 mg/dl, and/or Postprandial blood glucose ≥ 200 mg/dl) will be randomized in two arms. Participants in arm-1 will receive once daily insulin Glargine (12 units) plus once daily Glulisine (4 units) at breakfast/dinner, along with OHAs at stable dose and titrated optimally. Participants in the arm-2 will receive once daily premix analogue insulin (30/70) 16 units at breakfast/dinner, along with OHAs at stable dose and will be titrated as per the treatment algorithm.

During the randomization visit, the selected subjects after the run in period will be given a subject number and randomized between two arms.

Anthropometric measurements and vital sign will be taken. Concomitant medication and adverse events will be noted. Glucose meter, strips, Insulin and study diary will be dispensed. Training on Glucose meter usage, hypoglycemia, hyperglycemia symptoms, Insulin injection technique and dose titration technique will be done. Subjects will be instructed to maintain the record of dosing details in the patient diary. They will be given Diet and Exercise counselling. They will be asked to hand over the study diary and Insulin pen (empty or full) to the coordinator at each visit.

First three months will be an insulin dose titration period in which the subjects will be asked to visit the clinic at 12 weeks. Telephonic visit at week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 and 11. At week 4, and 8 investigator can have an unscheduled visit for training or insulin dispensing. During the telephonic visit subjects will be asked about concomitant medication and adverse events. During clinic visit at 12 weeks or unscheduled visit at week 4 or 8 anthropometric measurements, vital signs, concomitant medication and adverse event will be recorded. Glucometer strips, Insulin and study diary will be dispensed. The Insulin and study diary given during previous visit will be collected. The dose of Insulin will be titrated according to the algorithm given in appendix below with the 7 point SMBG done by the subject ±5 days before the following weeks 4, 8 & 12 and also insulin dose can be titrated by finger prick FBS and PPBS done at week 2, 6 and 10.

After 3 months, participants in arm-1 may undergo intensification to 2 injections of Glulisine if HbA1c is > 7% and/or 2-h postprandial glucose is >140 mg/dL. After 3 months, participants in arm-2 premix OD can be made BD if HbA1c is > 7% and/or 2-h postprandial glucose is >140 mg/dL despite effective titration of existing doses.

The next three months will be an insulin dose maintenance period in which the subjects will be asked to visit the clinic at 24 week. At week 16 and 20 telephonic visit or an unscheduled visit will be performed. During the telephonic visit they will be asked about concomitant medication and adverse events. During clinic visit at 24 weeks or unscheduled visit at week 16 or 20, anthropometric measurements, vital signs, concomitant medication and adverse event will be recorded. Glucometer strips, Insulin and study diary will be dispensed. The Insulin and study diary given during previous visit will be collected. The dose of Insulin, if needed will be titrated according to algorithm given in appendix below with the 7 point SMBG done by the subjects ±5 days before the following week 16, week 20 and week 24.

During the clinic visit at weeks 12 and 24, Medical history, Physical examination, laboratory investigations like blood glucose (fasting & 2hr after meal), HbA1c, Urea, Creatinine, Liver function test, Lipid profile, Urine albumin/creatinine ratio, urine pregnancy (if applicable) and ECG at week 24 will be done.

During the end of study visit at week 24 the subject will undergo medical examination, anthropometric measurements, vital signs, concomitant medication and adverse event will be recorded. The Insulin and study diary given during previous visit will be collected.

Subjects experiencing any hypoglycemia should inform the coordinator or the investigator over the phone and make an unscheduled visit. In case they experience adverse event should inform the coordinator or the investigator over the phone and make an unscheduled visit as per investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Insulin naïve men and women with T2DM on stable dose of 2 or 3 OHAs for at least 3 months.
2. Both men and women of age ≥ 18 and ≤ 65 years.
3. Have an HbA1c ≥ 7.5% and ≤ 10.5% with fasting blood glucose ≥ 150 mg/dl, and/or Postprandial blood glucose ≥ 200 mg/dl
4. Body mass index (BMI) ≤ 40 kg/m2.
5. Have given written informed consent to participate in this study in accordance with local regulations.
6. Subject must have access to telephone for calling into the clinical center as part of test product compliance.

Exclusion Criteria:

1. Type 1 diabetes
2. BMI > 40 kg/m2
3. Subject is being treated for severe active infection of any type
4. Have had more than one episode of severe hypoglycemia within 6 months prior to entry into the study.
5. Planned surgery in the next 6 months
6. Any event forecasted to require a temporary need to switch to insulin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1c | Baseline and 24 weeks
  To compare the change in HbA1c from baseline to week 24 between Glargine OD + Glulisine in comparison with Premixed insulin initiation in insulin naïve patients with T2DM

SECONDARY OUTCOMES:
Changes in Fasting Blood Glucose | Baseline and 24 weeks
  Effect of Glargine + Glulisine versus Premixed analogue Insulin in terms of changes in fasting blood glucose
Changes in postprandial blood glucose | Baseline and 24 weeks
  Effect of Glargine + Glulisine versus Premixed analogue Insulin in terms of changes in postprandial blood glucose
Changes in 7 point self monitored blood glucose profile | Baseline and 24 weeks
  Effect of Glargine + Glulisine versus Premixed analogue Insulin in terms of changes in 7 point self monitored blood glucose profile
Percentage reduction of HbA1c < 7% | Baseline and 24 weeks
  Effect of Glargine + Glulisine versus Premixed analogue Insulin in terms of percentage reduction of HbA1c < 7%
Changes in Insulin dose | Baseline and 24 weeks
  Effect of Glargine + Glulisine versus Premixed analogue Insulin in terms of changes in Insulin dose
Number of events of symptomatic hypoglycemia | Baseline and 24 weeks
  Effect of Glargine + Glulisine versus Premixed analogue Insulin in terms of number of events of symptomatic hypoglycemia
Number of events of severe hypoglycemia | Baseline and 24 weeks
  Effect of Glargine + Glulisine versus Premixed analogue Insulin in terms of number of events of severe hypoglycemia
Changes in weight | Baseline and 24 weeks
  Effect of Glargine + Glulisine versus Premixed analogue Insulin in terms of changes in Weight
Changes in Body mass index | Baseline and 24 weeks
  Effect of Glargine + Glulisine versus Premixed analogue Insulin in terms of changes in body mass index
Changes in blood pressure | Baseline and 24 weeks
  Effect of Glargine + Glulisine versus Premixed analogue Insulin in terms of changes in blood pressure
Number of participants treated related to adverse events | Baseline and 24 weeks
  Number of adverse event observed in both Glargine + Glulisine and Premixed analogue Insulin group will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Ambady Ramachandran, MD,Ph.D,D.Sc, Principal Investigator — President, India Diabetes Research Foundation
Locations (8):
- India (8):
  - Dr.Mallikarjnn Jali, Belagavi, Karnataka
  - Singhvi Health Centre, Chennai, Tamil Nadu
  - MedWay Hospitals, Chennai, Tamil Nadu
  - Kovai Diabetes Speciality Center and Hospital, Coimbatore, Tamil Nadu
  - Arthur Asirvatham Hospital, Madurai, Tamil Nadu
  - M.G.Diabetes Speciality and Research Center, Salem, Tamil Nadu
  - Ramana Maharishi Rangammal Hospital, Tiruvannamalai, Tamil Nadu
  - Trichy Diabetes Speciality Center (P) Ltd, Trichy, Tamil Nadu

IPD SHARING:
Plan to Share IPD: Undecided